CLINICAL TRIAL: NCT02628457
Title: Did MRI Appearance of Supraspinatus Muscle Atrophy Changes After Repair of All Kind of Rotator Cuff Tear?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CM Chungmu Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMH-2015-02
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Rotator Cuff Tear
Keywords: occupation ratio; pseudoatrophy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Mild Subgroup: patients with supraspinatus tendon retracted upto medial 1/3rd of humerus head and arthroscopic rotator cuff repair done by single row.
  Interventions: Procedure: arthroscopic rotator cuff repair
- Moderate Subgroup: patients with supraspinatus tendon retracted between medial 1/3rd of humerus head and glenoid,and arthroscopic rotator cuff repair done by single row.
  Interventions: Procedure: arthroscopic rotator cuff repair
- Severe subgroup: patients with supraspinatus tendon retracted beyond glenoid and arthroscopic rotator cuff repair done by single row
  Interventions: Procedure: arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: arthroscopic rotator cuff repair — arthroscopic rotator cuff repair done in all patients to check whether, surgery itself changes the appearance of muscle atrophy in the supraspinatus in all patients irrespective of size of preoperative tendon retraction

SUMMARY:
There are two purpose of this study, first is to find whether arthroscopic rotator cuff repair is changing the appearance of supraspinatus muscle atrophy in each and every patient. Second, is to find how much approximate change one can expect depending on age and tendon retraction

DETAILED DESCRIPTION:
Retrospective review of 209 patients having both preoperative and immediate postoperative MRI done. Both preoperative and immediate postoperative occupancy ratio calculated and from that change in occupancy ratio calculated for each and every patient. Patient were divided in two major group according to age that is <60 years and >60 years and 3 subgroups of mild, moderate and severe depending on preoperative supraspinatus tendon retraction on coronal view of MRI. Postoperative occupation ratio was compared with preoperative occupation ratio within the subgroups and change in occupation ratio was used for comparison between the subgroup. Change in occupation ratio was also used for comparison between 2 major groups

ELIGIBILITY:
Inclusion Criteria:

1. Patients with degenerative rotator cuff tear who underwent single-row arthroscopic rotator cuff repair in our hospital.
2. Patients with preoperative MRI and postoperative MRI within 1 week of surgery in our hospital.
3. Patients with minimum grade 1 supraspinatus atrophy in preoperative MRI.

Exclusion Criteria:

1. Patients with preoperative MRI from outside hospital.
2. Patients with isolated subscapularis tear.
3. Patients with previous operation on the same shoulder joint.
4. Patients with MRI images that were not usable due to poor quality or absence of appropriate Y-view.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 209 patients with degenerative rotator cuff tear who underwent single-row arthroscopic rotator cuff repair between March 2012 and April 2015 in CM hospital
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
change in supraspinatus muscle atrophy | within 1 week after surgery
  Supraspinatus muscle atrophy was measured and evaluated according to the Thomazeau classification. Stage 1: slight atrophy occupation ratio (1.00-0.60), Stage 2: moderate atrophy occupation ratio (0.60-0.40), Stage 3: Severe atrophy occupation ratio(<0.40). Both preoperative and immediate postoperative occupancy ratio calculated and from that change in occupancy ratio calculated for each and every patient.Postoperative occupation ratio was compared with preoperative occupation ratio within the groups and change in occupation ratio was used for comparison between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: sang-Hoon Lhee, MD PhD, Study Chair — President, CM general Hospital; Anant kumar Singh, Principal Investigator — arthroscopy fellow, CM general Hospital
Locations (1):
- Chungmu General Hopsital, Yeongdeungpo-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Sharing of data on the website is against the policy of IRB Korea